CLINICAL TRIAL: NCT05167305
Title: The Second COVID-19 Wave: Collateral Impact on Patients of Liver Disease-A Record Based Cross-Sectional Study.
Brief Title: The Second COVID-19 Wave: Collateral Impact on Patients of Liver Disease
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-COVID-07
Record Dates: First submitted 2021-12-17; First posted 2021-12-22 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- liver disease without COVID-19 infection-April-May 2019
  Interventions: Other: This is an observational study
- liver disease without COVID-19 infection -April- May 2021
  Interventions: Other: This is an observational study

INTERVENTIONS:
Other: This is an observational study — This is an observational study

SUMMARY:
Hospital record of the patients of liver disease admitted from April-May 2021 and April-May 2019 will be reviewed. Patients will be analyzed and compared for the demographic characteristics, severity of liver disease at time of admission and outcome in form of survival or mortality, liver transplantation rates in the two time periods and the subsequent 30 d and 90 day readmission rate.

Monitoring and assessment: Hospital records of all patients of liver disease needing admission during the April-May 2019 and 2021, but without active COVID-19 infection, will be reviewed. Patients will be analyzed and compared for the demographic characteristics, severity of liver disease at time of admission and outcome in form of survival or mortality, liver transplantation rates in the two time periods and 30 d and 90 d readmission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of liver disease requiring hospital admission

Exclusion Criteria:

1. Active COVID-19 infection at time of admission or acquiring during hospital stay.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of liver disease without COVID-19 infection admitted in the time period April- May 2021 and April-May 2019.
Sampling Method: Non-Probability Sample
Enrollment: 1316 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of in-hospital mortality rate of patients of liver disease admitted in April-May 2021 and April-May 2019. | Until discharge or death

SECONDARY OUTCOMES:
Comparison of 30 days readmission rate of patients of liver disease. | Day 30
Comparison of 31 to 90 days readmission rate of patients of liver disease. | Day 31-90
Comparison of liver transplantation rates in the two time periods i.e., April-May 2021 and April-May 2019. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No